CLINICAL TRIAL: NCT00246155
Title: A Prospective Study to Evaluate the Potential Effects on Function and Size in Back Muscle After Injection of Botulinum Toxin Type A (Dysport®) in the Treatment of Chronic Low Back Pain
Brief Title: Study on the Effects of Botulinum Toxin Type A on Back Muscle in Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-38-52120-103
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Low Back Pain
Keywords: chronic; muscular
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of this study is to analyse the changes in back muscle size and strength following use of Dysport®, and to establish whether there is any association between pain reduction and change in strength, in patients suffering from chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from muscular low back pain (between L-1 and S-1 level).
* Symptoms of more than six months duration.
* No benefit from previous treatments.
* Patient must present with bilaterally more than 2 active trigger points (TrPs) in the region of the low back musculature.
* CT scan or MRI examination of the lumbar spine was performed within the past year.
* Absence of significant pathology, such as bone fracture, nerve damage or severe psychiatric condition.

Exclusion Criteria:

* Constant or persistent severe pain due to nerve root compression or fibromyalgia.
* The patient has received surgery on the spine.
* Other musculoskeletal disabilities e.g. myasthenia gravis, or disorders of the neuromuscular junction.
* Any serious pathology, such as cancer, systemic inflammatory disease, vertebral fractures, neurological signs, spinal infection.
* Epidural injection of local anaesthetics and steroids within 12 weeks proceeding inclusion.
* Trigger point injection of local anaesthetics and steroid within 8 weeks proceeding inclusion.
* Pain associated with urinary tract infections, or gynaecological disorders.
* Bleeding disturbances or currently using coumarin derivatives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2005-01; Primary Completion 2005-07-01 (Actual); Study Completion 2005-07-01 (Actual)

PRIMARY OUTCOMES:
Pain reduction as assessed by the mean Visual Analogue Scale (VAS) during last 2 weeks. Assessments will be made at the initial time before injection and 1, 2, 3 months after injection.
Improvement in daily life activities and quality of life using the Oswestry Low Back Pain Questionnaire (OLBPQ), and Short Form-36 (SF-36). Assessments will be made at the initial time before injection and 1, 2, 3 months after injection.

SECONDARY OUTCOMES:
Changes of the total isometric lumbar extensor strength and separated angle using lumbar MedX machine.
Association between pain reduction and strength. Measurements will be performed at baseline, and 1, 2, 3 months after injection.
Change of the lumbar extensor muscular size in CT Measurement will be performed at baseline and 3 months after injection.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Wooridul Spine Hospital, Seoul, South Korea